CLINICAL TRIAL: NCT00888147
Title: Pilot Study: "Does Using a Fiber Containing Enteral Tube Feeding Formula Increase Constipation and the Use of Stool Softeners in Patients Undergoing Radiation Therapy and Have a Percutaneous Endoscopic Gastrostomy (PEG) Placed?"
Brief Title: Fiber Formula Study Among Radiation Oncology Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Lisa Epp, Home Enteral Nutrition Coordinator, Mayo Clinic
Other Study IDs: 08-005304
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2011-09-26 (Estimated); Status verified 2011-09

CONDITIONS: Constipation
Keywords: Tube feeding; Fiber; Constipation
MeSH Terms: conditions — Constipation | interventions — Proteins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fiber formula: This group will receive tube feeding formula that contains fiber.
  Interventions: Dietary Supplement: Fiber containing tube feeding formula

INTERVENTIONS:
Dietary Supplement: Fiber containing tube feeding formula — This group will be prescribed adequate calories, protein and fluid using a formula that contains fiber.
  Other Names: There is no brand name we are using. We will use the formula that best meets the patient calorie, protein and fluid needs.

SUMMARY:
During radiation treatment for head and neck cancer a large percentage of patients at Mayo Clinic Rochester develop the need for tube feeding to meet nutrition and hydration needs. These patients are usually taking pain medication along with a stool softener or laxative. Currently, when these patients get a feeding tube it is our standard practice to choose a fiber-free enteral tube feeding formula as to not worsen their constipation. Currently, there are no guidelines as to which patients are good candidates for fiber containing enteral tube feeding formulas. The investigators hope this study will help determine if fiber containing enteral tube feeding formulas can be used for patients undergoing radiation for head and neck cancer without increasing rates of constipation or increasing use of stool softeners/laxatives.

Hypothesis: Participants enrolled in the study will not have increased rates of constipation on fiber-containing enteral tube feeding formula compared to historical standards on fiber-free formula.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of: 1) lip/oral cavity 2) pharynx 3) larynx 4) nasal cavity/paranasal sinus 5) salivary gland 6) Thyroid according to AJCC cancer staging manual 6th edition 2002
* Current radiation therapy or starting radiation therapy in the next 2 weeks
* Patient must have a gastrostomy tube

Exclusion Criteria:

* Jejunostomy tube
* Diagnosis of Irritable Bowel Syndrome (abdominal pain and diarrhea or constipation lasting at least three months in one year)
* Short bowel (A patient is generally considered to have short bowel syndrome when less than 100 to 150 centimeters of functioning small bowel remains)
* Body max index (BMI) <18.5kg/m2
* Gastroparesis (when the stomach retains food for longer than normal periods). This must be diagnosed with a gastric emptying study.
* Use of Metoclopramide
* Receiving 5-FU chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These participants have head and neck cancer, are undergoing radiaiton therapy and will have a percutaneous endoscopic gastrostomy (PEG) placed.
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2009-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Whether each patient gets constipated. | Weekly for 2 weeks

SECONDARY OUTCOMES:
Whether the amount of stool softeners/laxatives increases in comparison to the original recommended regimen, for each individual patient. | Weekly for 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa M Epp, BS, Principal Investigator — Mayo Clinic; Yolanda I Garces, MD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States